CLINICAL TRIAL: NCT04756674
Title: Investigating the Impact of COVID-19 Infection on Skeletal Muscle
Brief Title: The Impact of Covid-19 on Skeletal Muscle
Status: Withdrawn | Type: Observational
Why Stopped: Failure to recruit due to high use of anticoagulants in COVID-19 patients and rapid declining rates of COVID-19 thanks to the vaccine implementation
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 20065; Sponsor ID: 20065 (Other: University of Nottingham)
Record Dates: First submitted 2020-11-02; First posted 2021-02-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Muscle Loss; Mitochondrial Alteration
MeSH Terms: conditions — COVID-19; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: Non-Covid -19 associated community acquired pneumonia with oxygen therapy required.
  n=12
  Interventions: Other: No intervetion will be used
- Oxygen Therapy: Confirmed COVID-19 infection via PCR swab, with a new oxygen therapy requirement. NB the researchers will not be involved in the clinical decision of if the participant requires oxygen, this will be the clinical-teams decision.
  n=12
  Interventions: Other: No intervetion will be used
- Non-Invasive ventilation therapy: Confirmed COVID-19 infection via PCR Swab, with a clinical need for non-invasive ventilation.
  NB the researchers will not be involved in the clinical decision if the participant requires non-invasive ventilation, this will be the clinical-teams decision.
  n=12
  Interventions: Other: No intervetion will be used

INTERVENTIONS:
Other: No intervetion will be used — No intervention will be used

SUMMARY:
With the recent worldwide outbreak of the COVID-19 infection and the huge impact it has had upon lives in the UK, it is key to increase knowledge on the impact of the virus on the body. Certain aspects of the virus' characteristics are also poorly understood: The reason behind the variation in response between individuals, and the long-term impacts of infection upon the body. It is already known from previous research that muscle-health plays an important role in health, with other illnesses known to have an impact upon muscle health. A large number of studies have investigated the relationship between muscle and health, with an increasing focus upon the impact upon the mitochondria within the muscle cells. Mitochondria are the energy-producing component of a cell and are vital not just for the muscle-cells but for the body as a whole.

The researchers hope that by investigating the impact of COVID-19 infection upon human skeletal muscle, the question of why individuals have different responses to the infection and the mechanism of the longer-term impact of infection can be answered. This added knowledge will then, hopefully, be able to guide therapy targets in the future.

DETAILED DESCRIPTION:
Since the outbreak of the COVID-19 pandemic worldwide, there have been over 50,000 deaths and over 1million infections in the UK alone. It has been widely reported that infection with COVID-19 leads to large variation between individuals, a large number appear asymptomatic or mild flu-like symptoms compared to a percentage requiring intensive care support and for some, the infection is ultimately fatal. The reason behind this variation is not yet fully understood.

With COVID-19 likely to have a lasting impact within the UK and on the NHS, any research that improves our knowledge upon the effect of the infection has the possibility to improve therapy targets and hopefully improve patient outcomes.

With how novel the COVID-19 pathogen is, little is currently known about the potential long-term impacts of infection upon individuals. There are currently many reports of longer-term syndromes following infection with COVID-19 including loss of smell and myalgia. The researchers hope that investigating the impact upon patients over the 12-months following their infection will gather information on the long-term impacts and potentially find evidence of the reason for these longer-term symptoms.

With skeletal muscle being one of the largest components of the human body, any impact upon its function is likely to have a significant impact upon an individual. With it being vital for not only locomotion but also in energy production for the body. The researchers hypothesize that changes within the skeletal muscle may account for some of the impacts of COVID-19 infection. The investigators hope that by investigating changes in muscle structure, muscle mitochondrial function, and neurological supply to the muscle they can identify a future therapy target to improve outcomes from COVID-19 infection.

To investigate this, this study plans to recruit participants with confirmed COVID-19 infection requiring varying levels of oxygen support (Oxygen therapy only n=12, Non-invasive ventilation n=12) and a control group of non-covid community-acquired pneumonia requiring oxygen therapy (n=12).

All groups will undergo the same investigations, and no interventions will form part of the study. Investigations will be carried out at 24-72hours of acute hospital admission, with follow-up assessments at 6-months and 12-months post-discharge.

The assessments performed will include: muscle biopsy of the vastus lateralis muscle, an ultrasound scan of the vastus lateralis muscle, voluntary and stimulated iEMG of VL, and hand-grip strength analysis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection as confirmed by PCR swab, or being treated for non-COVID-19 community acquired pneumonia
* A minimum of oxygen treatment required for 24hours.
* Capacity to give informed and written consent

Exclusion Criteria:

* A BMI <16.5 or >35 kg/m2
* Active cardiovascular disease:

Significant arrhythmia

Recent acute coronary event

* Cerebrovascular disease:

Recent stroke

* Respiratory disease including:

Pulmonary hypertension

Significant COPD

Uncontrolled asthma

* Clotting dysfunction or current use of anticoagulants (eg Warfarin/Clopidogrel/ Rivaroxaban)
* Significant musculoskeletal or neurological disorders

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of individuals being treated for COVID-19 infection with a minimum of oxygen therapy.
  Control population of individuals being treated for non-COVID-19 community acquired pneumonia requiring oxygen therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The difference in mitochondrial function between COVID-19 infection and control group | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Assessment of skeletal muscle mitochondrial oxidative phosphorylation rate between COVID-19 associated illness and Control group (non-covid community-acquired pneumonia).
  This will be assessed by measuring oxygen consumption using a high-resolution respirometer and expressed as a ratio of maximal rate.
The difference in mitochondrial function between levels of ventilation support required in COVID-19 patients | each of the 3 time points assessed: the acute admission, as well as in the recovery phases - 6 month and 12 month follow up
  Assessment of skeletal muscle mitochondrial oxidative phosphorylation rate assessed using high-resolution respirometer between the 2 groups of ventilatory support in COVID-19 patients (Oxygen only support, non-invasive ventilation). Expressed as a ratio of maximal oxygen consumption.
The changes in mitochondrial function during the recovery period from COVID-19 | Comparison over the 3 time periods: acute admission, 6month and 12 month follow up
  Assessment of skeletal muscle mitochondrial oxidative phosphorylation rate using high-resolution respirometer expressed as a percentage change over the time period in each group

SECONDARY OUTCOMES:
The difference in muscle macroscopic structure between the groups | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Ultrasound will allow the research group to provide an estimate of vastus lateralis size (mm3).
  This will be compared between the 3 groups.
The difference in muscle macroscopic structure between the groups | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Ultrasound will allow the research group to provide an estimate of fascicle length (mm) between the 3 groups.
The difference in muscle macroscopic structure between the groups | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Ultrasound will allow the research group to provide an estimate of fascicle angle (degrees) between the 3 groups.
Difference in the neurological supply of skeletal muscle | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Measuring iEMG activity from voluntary and involuntary contractions will allow a detailed examination of the nerve-muscle relationship assessed by nerve firing rate (hz)
Difference in the neurological supply of skeletal muscle | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Measuring iEMG activity from voluntary and involuntary contractions will allow a detailed examination of the nerve-muscle relationship encompassing the neuromuscular junction transmission stability (assessed using MUP (uv.ms)
Difference in the neurological supply of skeletal muscle | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  Measuring iEMG activity from voluntary and involuntary contractions will allow a detailed examination of the nerve-muscle relationship allowing us to assess nerve conduction time (ms)
Difference in muscle function | This will be assessed in each of the 3 time points: the acute admission assessment, as well as in the recovery period of 6-month and 12-month follow up
  This will be analysed according to handgrip strength performance (measured in kg)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Phillips, BSc PhD, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided